CLINICAL TRIAL: NCT05999097
Title: To Study the Clinical Effect of SC-FOS Prebiotics in Enteral Diet vs. Standard Enteral Diet on Clinical Characteristics of Patients With Polycystic Ovary Syndrome According to the Rotterdam Classification in Chihuahua, Chihuahua. A Randomized Single-Blind Clinical Trial
Brief Title: To Study the Effect of SC-FOS Prebiotics in Women With Polycystic Ovary Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Autonoma de Chihuahua (Other)
Responsible Party: Principal Investigator, Carolina Martínez Loya, MD, Medical Doctor, Universidad Autonoma de Chihuahua
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 030C-06/23
Record Dates: First submitted 2023-08-11; First posted 2023-08-21 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-02

CONDITIONS: Polycystic Ovary Syndrome
Keywords: Polycystic Ovary Syndrome; Prebiotics; Enteral Diet; Clinical Manifestations; SC-FOS
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Prospective study, randomized single blind clinical trial
Who Masked: Participant
Masking Description: Single (Participant)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short Chain Fructooligosaccharides Group (Experimental): This group will receive Short-Chain Fructooligosaccharides at a dose of 12 gr. every 24 hours for 10 days, diluted in 250 ml
  Interventions: Dietary Supplement: Short Chain Fructooligosaccharides
- Placebo Group (Placebo Comparator): This group will receive Corn Starch as a Placebo control 12 gr. every 24 hours for 10 days, diluted in 250 ml
  Interventions: Dietary Supplement: Placebo Group

INTERVENTIONS:
Dietary Supplement: Short Chain Fructooligosaccharides — The intervention will receive Short-Chain Fructooligosaccharides at a dose of 12 gr. every 24 hours diluted in 250 ml of water.
  Other Names: Prebiotics
  Arms: Short Chain Fructooligosaccharides Group
Dietary Supplement: Placebo Group — This group will receive 12 g of corn starch as a control group.
  Other Names: Placebo
  Arms: Placebo Group

SUMMARY:
The purpose of this study is to determine if there is a difference in the clinical characteristics of patients with polycystic ovary syndrome after the administration of SC-FOS in the enteral diet compared to patients with a standard diet.

DETAILED DESCRIPTION:
The protocol will be discussed with the patients and/or relatives of the patients, who will understand the consequences and advantages of the study and will thus sign the consent.

Once informed consent has been obtained, the group to which each patient belongs will be randomly assigned.

Patients will be selected according to the inclusion and exclusion criteria of the population diagnosed with PCOS with useful enteral route for random assignment into two groups, one will be administered short-chain Fructooligosaccharides at a dose of 12 g every 24 hours, another group will be given saline as a placebo to the enteral diet every 24 hours for 10 days. Patients should take the solution on an empty stomach.

Once the type of intervention has been determined, the patient will be given the suspensions corresponding to group 1 or placebo, with vials in which the content cannot be visualized, numbered according to the sheet obtained by the corresponding randomization. The initial evaluation will be completed with all the clinical characteristics to be evaluated.

The patient will be told that every 24 hours he must take 1 suspension on an empty stomach, which will be prepared at a rate of 12 grams of SC-FOS in 15 cc of saline solution for the prebiotic preparation vs 15 cc of saline solution for the placebo group. The solution will be administered enterally for 10 consecutive days at a single dose per day, and a reassessment will be made on the seventh day of the clinical characteristics of the patients, to compare and evaluate the results.

ELIGIBILITY:
Inclusion Criteria:

* Female sex
* Age 18 to 65 years
* Polycystic Ovary Syndrome diagnosed by specialist
* Useful enteral feeding

Exclusion Criteria:

* Pregnancy
* Diabetes mellitus
* Risk of intestinal perforation

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-02 (Estimated); Primary Completion 2025-05-10 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
Score of Bristol Scale | 10 days
  Score obtained by Stool Consistency Bristol Scale:
  This scale consist in seven types of stool:
  Type 1: Separate hard lumps, like nuts (difficult to pass) Type 2: Sausage-shaped, but lumpy Type 3: Like a sausage but with cracks on its surface Type 4: Like a sausage or snake, smooth and soft (average stool) Type 5: Soft blobs with clear cut edges Type 6: Fluffy pieces with ragged edges, a mushy stool (diarrhea) Type 7: Watery, no solid pieces, entirely liquid (diarrhea)
Score Short Form Health Survey (SF-36) | 10 days
  Short Form Health Survey (SF-36) is a measure of health-related quality-of-life:
  It comprises 36 questions that cover eight domains of health
  1. Limitations in physical activities because of health problems.
  2. Limitations in social activities because of physical or emotional problems
  3. Limitations in usual role activities because of physical health problems
  4. Bodily pain
  5. General mental health (psychological distress and well-being)
  6. Limitations in usual role activities because of emotional problems
  7. Vitality (energy and fatigue)
  8. General health perceptions

CONTACTS AND LOCATIONS:
Overall Officials: Luis B Enríquez-Sánchez, Study Director — Universidad Autonoma de Chihuahua
Locations (1):
- Hospital Central del Estado de Chihuahua, Chihuahua City, Mexico

IPD SHARING:
Plan to Share IPD: Yes
The data obtained from this research study will be available if requested once the study is finalized.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data will be available for up to five years since completion of the study.
Access Criteria: The request for the data will be by e-mail